CLINICAL TRIAL: NCT00849264
Title: a Randomized Controlled Study of Surgical Comprehensive Treatment for Different Types of Tumor Thrombi in the Portal Vein for Hepatocellular Carcinoma Patients
Brief Title: Comprehensive Treatment for Different Types of Tumor Thrombi in the Portal Vein for Hepatocellular Carcinoma Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Hepatobiliary Surgery Hospital (Other)
Responsible Party: Principal Investigator, ShenFeng, vice president of the Eastern Hepatobiliary Surgery Hospotal, Eastern Hepatobiliary Surgery Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EHBH-RCT-2008-004
Record Dates: First submitted 2009-02-19; First posted 2009-02-23 (Estimated); Last update posted 2016-04-01 (Estimated); Status verified 2016-03

CONDITIONS: Hepatocellular Carcinoma; Portal Vein Tumor Thrombus
Keywords: hepatocellular carcinoma; portal vein tumor thrombus; surgical comprehensive treatment
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Drug Therapy; endostar protein; Therapeutics; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A (Experimental): PLC patients with PVTT underwent hepatectomy and portal thrombectomy followed by portal vein chemotherapy with endostar
  Interventions: Drug: chemotherapy with endostar
- B (Active Comparator): PLC patients with PVTT underwent hepatectomy and portal thrombectomy followed by portal vein chemotherapy with CBP and 5-FU
  Interventions: Drug: treatment with CBP and 5-FU
- C (Experimental): PLC patients with PVTT underwent hepatectomy and portal thrombectomy followed by portal vein chemotherapy with endostar, CBP and 5-FU
  Interventions: Drug: treatment with endostar, CBP and 5-FU

INTERVENTIONS:
Drug: chemotherapy with endostar — 15mg/d×14d
  Other Names: chemotherapy with endostar group
  Arms: A
Drug: treatment with CBP and 5-FU — CBP 300mg/d×2d，5-FU 1000mg/d×5d
  Other Names: treatment with CBP and 5-FU group
  Arms: B
Drug: treatment with endostar, CBP and 5-FU — CBP 300mg/d×2d，5-FU 1000mg/d×5d ，Endostar 15mg/d×14d
  Other Names: endostar, CBP and 5-FU group
  Arms: C

SUMMARY:
This study is working to evaluate the surgical comprehensive treatment for different types of tumor thrombi in the portal vein for hepatocellular carcinoma patients, to establish a standardized, unified, effective therapeutic program.

DETAILED DESCRIPTION:
Primary liver cancer (PLC) has a great tendency to invade portal vein intravascularly, results in the formation of portal vein tumor thrombus (PVTT), which is a crucial factor that can worsen the prognosis of patients with PLC.

In clinical, various treatments have been applied to improve this short-term prognosis, but there was no identical indication for treatment of PLC patients with different PVTT.

The objective of this study is to evaluate the surgical comprehensive treatment for different types of tumor thrombi in the portal vein for hepatocellular carcinoma patients, to establish a standardized, unified, effective therapeutic program.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients > 30 years and <=60 years of age.
* with a clinical diagnosis of primary liver cancer with PVTT, without any adjuvant therapy.
* resectable tumors in the liver.
* PVTT type for II or III (based on the PVTT type system established by our groups), confirmed through pre-operative imaging and pathologic examination.
* liver function grade A or B of the Child-Pugh classification.
* No dysfunction in major organs; Blood routine, kidney function, cardiac function and lung function are basically normal. Hb ≥95g/L,WBC ≥3.000 cells/mm³,platelets ≥80.000 cells/mm³.
* Patients who can understand this trial and have signed information consent.

Exclusion Criteria:

* have had an allergic reaction following iodine or chemotherapeutic drugs.
* with extrahepatic metastasis.
* Patients with apparent cardiac, pulmonary, cerebral and renal dysfunction,which may affect the treatment of liver cancer.
* liver function:Child C.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
overall survival | 2010

SECONDARY OUTCOMES:
disease-free survival | 1,2 and 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Feng Shen, M.D., Study Chair — Eastern Hepatobiliary Surgery Hospital, Second Military Medical University
Locations (1):
- Eastern hepatobilliary surgery hospital, Shanghai, Shanghai Municipality, China